CLINICAL TRIAL: NCT07221643
Title: Carotenoids in the Skin and Immune Aging: a Pilot Observational Study
Brief Title: Carotenoids in the Skin and Immune Aging
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anne Chang, Professor of Dermatology, Stanford University
Other Study IDs: 80982
Record Dates: First submitted 2025-09-30; First posted 2025-10-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: No Condition; Skin Carotenoids and Immune-aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young adult: Participants are 18 to 30 years old.
- Older adult: Participants are over 65 years old.

SUMMARY:
This study aims to examine the connection between the level of carotenoids in the skin and a number of immune related health parameters.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Age 18-30 years OR 65 years and older
* Healthy individuals without uncontrolled medical conditions (over the counter inhaled and topical steroids allowed)
* Fiitzpatrick I-VI (all skin types)

Exclusion Criteria:

* Pregnant or breastfeeding
* uncontrolled medical conditions
* Skin conditions on the upper extremity that would interfere with skin measurements of carotenoid levels such as active atopic dermatitis or psoriasis
* Concurrent use of medications that affect the immune system, within 4 weeks of enrollment (eg. prednisone, biologics, methotrexate, rapamycin, prescription topical steroids, prescription inhaled steroids, others)
* Unable to follow study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals who are either between 18 to 30 years old or over 65 years old.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Skin carotenoid levels and skin aging features | one day
  We will assess the skin carotenoid levels' correlation with skin aging features, such as wrinkles, fine lines, and age spots.

SECONDARY OUTCOMES:
Skin carotenoid levels and biomarkers of aging | one day
  We will assess the skin carotenoid levels' correlation with biomarkers associated with aging, such as C-reactive protein, telomere length, telomerase activity etc.
Skin carotenoid levels and self-reported perception of health | 2 weeks
  We will assess the skin carotenoid levels' correlation with self reported scores on general health and health beliefs, incidence of respiratory, gut and skin allergy symptoms, and sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Health - General Dermatology Clinic, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No